CLINICAL TRIAL: NCT02169466
Title: Pharmacokinetic-pharmacodynamic Interaction Between Three Different Single Doses of BIA 9-1067 and a Single-dose of Controlled-release 100/25 mg Levodopa/Benserazide: a Double-blind, Randomized, Four-way Crossover, Placebo-controlled Study in Healthy Male Subjects
Brief Title: Pharmacokinetic-pharmacodynamic Interaction Between Three Different Single Doses of BIA 9-1067 and a Single-dose of Controlled-release 100/25 mg Levodopa/Benserazide
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIA-91067-109
Record Dates: First submitted 2012-01-20; First posted 2014-06-23 (Estimated); Results first posted 2015-11-03 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-10

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's disease (PD); Opicapone; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental): Period 1: BIA 9-1067 25 mg Period 2: BIA 9-1067 50 mg Period 3: BIA 9-1067 100 mg Period 4: Placebo
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Madopar® HBS (Single-dose of controlled-release levodopa/benserazide 100/25 mg: 1 capsule of Madopar® HBS.)
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Madopar® HBS
- Group 2 (Experimental): Period 1: BIA 9-1067 50 mg Period 2: BIA 9-1067 100 mg Period 3: Placebo Period 4: BIA 9-1067 25 mg
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Madopar® HBS (Single-dose of controlled-release levodopa/benserazide 100/25 mg: 1 capsule of Madopar® HBS.)
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Madopar® HBS
- Group 3 (Experimental): Period 1: BIA 9-1067 100 mg Period 2: Placebo Period 3: BIA 9-1067 25 mg Period 4: BIA 9-1067 50 mg
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Madopar® HBS (Single-dose of controlled-release levodopa/benserazide 100/25 mg: 1 capsule of Madopar® HBS.)
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Madopar® HBS
- Group 4 (Experimental): Period 1: Placebo Period 2: BIA 9-1067 25 mg Period 3: BIA 9-1067 50 mg Period 4: BIA 9-1067 100 mg
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Madopar® HBS (Single-dose of controlled-release levodopa/benserazide 100/25 mg: 1 capsule of Madopar® HBS.)
  Interventions: Drug: BIA 9-1067; Drug: Placebo; Drug: Madopar® HBS

INTERVENTIONS:
Drug: BIA 9-1067 — OPC, Opicapone
  Other Names: OPC, Opicapone
Drug: Placebo — PLC, Placebo
  Other Names: PLC, Placebo
Drug: Madopar® HBS — controlled-release levodopa 100 mg/benserazide 25 mg

SUMMARY:
To investigate the effect of three single oral doses of BIA 9-1067 (25 mg, 50 mg and 100 mg) on the levodopa pharmacokinetics when administered in combination with a single-dose of controlled-release levodopa 100 mg/benserazide 25 mg (Madopar HBS).

DETAILED DESCRIPTION:
Single centre, double-blind, randomized, placebo-controlled, crossover study with four consecutive single-dose treatment periods. The washout period between doses was to be at least10 days. On each treatment period (25, 50 and 100 mg BIA 9-1067 or placebo), after completion of pre-dose assessments, BIA 9-1067-Placebo was to be administered concomitantly with the dose of Madopar HBS; post-dose assessments were to be completed and subjects were to be discharged 72 h post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, complete neurological examination and 12-lead ECG.
* Subjects who had clinical laboratory test results that were clinically acceptable at screening and admission to first treatment period.
* Subjects who had negative tests for hepatitis B surface antigen (HBsAg), anti-hepatitis C antibodies (HCV Ab), and Human immunodeficiency viruses -1 and -2 antibodies (HIV-1 and HIV-2 Ab) at screening.
* Subjects who had/were negative for drugs of abuse at screening and admission to each treatment period.
* Subjects who were non-smokers or who smoked ≤10 cigarettes or equivalent per day.
* Subjects who were able and willing to give written informed consent.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria, or
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity.
* Subjects who had a history of glaucoma.
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 21 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening or first admission.
* Subjects who had acute gastrointestinal symptoms at the time of screening or first admission (e.g., nausea, vomiting, diarrhoea, heartburn).
* Subjects who used medicines within 2 weeks of first admission that, in the opinion of the investigator, may affect the safety or other study assessments.
* Subjects who used any investigational drug or participated in any clinical trial within 2 months of their first admission.
* Subjects who donated or received any blood or blood products within the previous 2 months prior to screening.
* Subjects who were vegetarians, vegans or have medical dietary restrictions.
* Subjects who could not communicate reliably with the investigator.
* Subjects who were unlikely to co-operate with the requirements of the study.
* Subjects who were unwilling or unable to give written informed consent.
* Subjects who were BIAL - Portela & Cª, SA employees.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2009-01; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BIAL - Portela & Cª - Human Pharmacology Unit (UFH), S. Mamede Do Coronado, Trofa, Portugal

RESULTS

PARTICIPANT FLOW:
Groups:
- BIA 9-1067: 25, 50, 100, Placebo: Period 1: BIA 9-1067 25 mg Period 2: BIA 9-1067 50 mg Period 3: BIA 9-1067 100 mg Period 4: Placebo
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Madopar® HBS (Single-dose of controlled-release levodopa/benserazide 100/25 mg: 1 capsule of Madopar® HBS.)
  BIA 9-1067: OPC, Opicapone
  Placebo: PLC, Placebo
  Madopar® HBS: controlled-release levodopa 100 mg/benserazide 25 mg
- BIA 9-1067: 50, 100, Placebo, 25: Period 1: BIA 9-1067 50 mg Period 2: BIA 9-1067 100 mg Period 3: Placebo Period 4: BIA 9-1067 25 mg
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Madopar® HBS (Single-dose of controlled-release levodopa/benserazide 100/25 mg: 1 capsule of Madopar® HBS.)
  BIA 9-1067: OPC, Opicapone
  Placebo: PLC, Placebo
  Madopar® HBS: controlled-release levodopa 100 mg/benserazide 25 mg
- BIA 9-1067: 100, Placebo, 25, 50: Period 1: BIA 9-1067 100 mg Period 2: Placebo Period 3: BIA 9-1067 25 mg Period 4: BIA 9-1067 50 mg
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Madopar® HBS (Single-dose of controlled-release levodopa/benserazide 100/25 mg: 1 capsule of Madopar® HBS.)
  BIA 9-1067: OPC, Opicapone
  Placebo: PLC, Placebo
  Madopar® HBS: controlled-release levodopa 100 mg/benserazide 25 mg
- BIA 9-1067: Placebo, 25, 50, 100: Period 1: Placebo Period 2: BIA 9-1067 25 mg Period 3: BIA 9-1067 50 mg Period 4: BIA 9-1067 100 mg
  BIA 9-1067/Placebo was to be administered concomitantly with the dose of Madopar® HBS (Single-dose of controlled-release levodopa/benserazide 100/25 mg: 1 capsule of Madopar® HBS.)
  BIA 9-1067: OPC, Opicapone
  Placebo: PLC, Placebo
  Madopar® HBS: controlled-release levodopa 100 mg/benserazide 25 mg
Period: Overall Study
Arm/Group | BIA 9-1067: 25, 50, 100, Placebo | BIA 9-1067: 50, 100, Placebo, 25 | BIA 9-1067: 100, Placebo, 25, 50 | BIA 9-1067: Placebo, 25, 50, 100
Started | 6 | 6 | 5 | 5
25 mg BIA 9-1067 | 6 | 5 | 5 | 5
50 mg BIA 9-1067 | 6 | 6 | 5 | 5
100 mg BIA 9-1067 | 6 | 6 | 5 | 5
Placebo | 5 | 6 | 5 | 5
Completed | 5 | 5 | 5 | 5
Not Completed | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIA 9-1067: 25, 50, 100, Placebo | BIA 9-1067: 50, 100, Placebo, 25 | BIA 9-1067: 100, Placebo, 25, 50 | BIA 9-1067: Placebo, 25, 50, 100 | Total
Number analyzed (Participants) | 6 | 6 | 5 | 5 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 5 | 5 | 22
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 5 | 5 | 22

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Plasma Concentration of Levodopa
Description: Primary pharmacokinetic parameter: Levodopa maximum observed plasma concentration (Cmax) (ng/mL)
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 h post-dose.
Population: According to the protocol, the "pharmacokinetic population" should include all subjects who had valid data for all treatment periods.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- BIA 9-1067 25 mg: BIA 9-1067 25 mg OPC Opicapone Of the initialy enrolled 21 subjects, 1 subject was not considered for the accountability as he was withdrawn from study participation
- BIA 9-1067 50 mg: BIA 9-1067 50 mg OPC Opicapone
- BIA 9-1067 100 mg: BIA 9-1067 100 mg OPC Opicapone
- Placebo: Placebo, PLC Of the initialy enrolled 21 subjects, 1 subject was not considered for the accountability as he was withdrawn from study participation
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
ng/mL | 314 (110) | 266 (77.5) | 263 (94.9) | 260 (119)

2. Primary Outcome: AUC0-t - Area Under the Plasma Concentration-time Curve
Description: Primary pharmacokinetic parameter: Area under the plasma concentration-time curve for levodopa
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 h post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Groups:
- BIA 9-1067 25 mg: BIA 9-1067 25 mg OPC Opicapone Of the initially enrolled 21 subjects, 1 subject was not considered for the accountability as he was withdrawn from study participation
- Placebo: Placebo, PLC Of the initially enrolled 21 subjects, 1 subject was not considered for the accountability as he was withdrawn from study participation
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
ng.h/mL | 1084 (398) | 1064 (365) | 1140 (592) | 933 (422)

3. Primary Outcome: AUC0-∞ - AUC From Time Zero to Infinity
Description: Primary pharmacokinetic parameter: Area under the plasma concentration-time curve from time zero to infinity for levodopa
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 h post-dose.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Number analyzed (Participants) | 19 | 20 | 19 | 19
ng.h/mL | 1190 (441) | 1181 (373) | 1326 (604) | 1086 (380)

4. Primary Outcome: Tmax - Time to Cmax
Description: Primary pharmacokinetic parameter: tmax - time to Cmax
Time Frame: pre-dose, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48 and 72 h post-dose.
Population: as for outcome 1
Measure: Mean (Full Range); unit: hours
Groups:
- BIA 9-1067 25 mg: BIA 9-1067 25 mg OPC Opicapone
- Placebo: Placebo, PLC
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Number analyzed (Participants) | 20 | 20 | 20 | 20
hours | 2.50 [1.0 to 4.0] | 2.50 [1.0 to 4.0] | 2.00 [1.0 to 6.0] | 2.00 [1.0 to 4.0]

ADVERSE EVENTS:
Time Frame: Just before drug administration until 72 h post-dose
Arm/Group | BIA 9-1067 25 mg | BIA 9-1067 50 mg | BIA 9-1067 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/22 | 0/22 | 0/21
Other Adverse Events (participants affected / at risk) | 2/21 | 4/22 | 3/22 | 2/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 25 mg (N=21) | BIA 9-1067 50 mg (N=22) | BIA 9-1067 100 mg (N=22) | Placebo (N=21)
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other